CLINICAL TRIAL: NCT03215602
Title: EXercise as TReatment for osteoArthritis
Acronym: EXTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Collaborators: The Danish Rheumatism Association (Other); Region Zealand (Other); Naestved Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Pætur Mikal Holm, PhD fellow, Slagelse Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJ-517
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; exercise; quadriceps; strength; activities of daily living; treatment outcome
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity | interventions — Educational Status; Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel group, assessor- and patient blinded randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One blinded outcome assessor (physiotherapists) will perform measurements of muscle strength, functional capacity and pain sensitization. The MRI scans will be performed by blinded radiologists. Patients in both groups will be blinded for parallel group assignments. Statistical analysis will be performed by a blinded statistician and a blinded interpretation of the results will be performed before breaking the randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEMEX and education + strength training (Experimental): Participants will undergo 12 weeks of twice weekly exercise. Each exercise session will last for 70-90 min. and will consist of 1 hour of specific exercises to optimize sensorimotor control and achieve compensatory functional stability performed in a multiple-joint weight-bearing specific manner. The final part of the session will consist of focused knee extensor strength training performed in gym machines (knee extension & leg-press) in a combination of low-load fatiguing exercises (knee-extension) followed by high-load exercises (leg-press).
  Additionally, participants will receive 2 educational sessions, which include disease- and exercise specific counseling.
  Interventions: Other: NEMEX and education + strength training
- NEMEX and education (Active Comparator): Participants will undergo 12 weeks of twice weekly exercise. Each exercise session will last for approximately 60 min. and will consist of 1 hour of specific exercises to optimize sensorimotor control and achieve compensatory functional stability performed in a multiple-joint weight-bearing specific manner.
  Additionally, participants will receive 2 educational sessions, which include disease- and exercise specific counseling.
  Interventions: Other: NEMEX and education

INTERVENTIONS:
Other: NEMEX and education + strength training — Optimizing sensorimotor control and achieving functional stability. Increasing knee extensor muscle strength. Teaching everyday disease management.
  Other Names: GLA:D + strength training
  Arms: NEMEX and education + strength training
Other: NEMEX and education — Optimizing sensorimotor control and achieving functional stability. Teaching everyday disease management.
  Other Names: GLA:D
  Arms: NEMEX and education

SUMMARY:
Osteoarthritis (OA) of the knee is a chronic musculoskeletal disease, and a major cause of pain and disability worldwide. Exercise has previously demonstrated good effect in alleviating OA symptoms. However, optimal exercise modes in OA are currently unknown.

This study seeks to evaluate the effects of supplementary focused, knee extensor strength training in addition to neuromuscular exercise (NEMEX) and education in people with OA of the knee as performed in Good Life with osteoArthritis in Denmark (GLA:D ᵀᴹ).

Through a randomized design, study participants will either be allocated to 12 weeks (twice weekly) of NEMEX and education or 12 weeks (twice weekly) of NEMEX and education and focused, knee extensor strength training.

The primary outcome measurement for this study is the Knee injury and Osteoarthritis Outcome Score, subscale Activities of Daily Living (KOOS-ADL), which is a self-reported questionnaire on daily life activities. Other outcomes include parameters of maximal muscle strength and muscle power, muscle imaging, physical function, pain and self-reported health status.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most prevalent musculoskeletal diseases worldwide. In Denmark, it is estimated that approximately 900.000 people, or 1 out of 5 residents are suffering from OA in one or more joints. The annual socio-economic costs (treatment and loss of labour) as a direct consequence of OA in Denmark are estimated to 11.5 billion "Danish kroner" (DKK).

Osteoarthritis of the knee is the most frequently reported and disabling OA subgroup and is mainly reported in middle-aged adults (≥40 years) with an increasing prevalence with increasing age. Knee osteoarthritis is associated with knee pain, loss of lower limb muscle strength, activity limitations and reduced quality of life. Moreover, pain sensitization, i.e. increased responsiveness of nociceptive neurons, is another mechanism involved in pain and disability in knee-OA and may contribute to the frequently reported disparities between pain symptoms and radiographic signs of structural damage.

The current non-surgical treatment recommendations in Denmark as well as internationally include offering one or more of: Patient education, dietary advice, weight loss counselling and exercise. Exercise has proven to be a potent stimulus to improve function, and general quality of life in people with knee-OA. Moreover, exercise has been shown to reduce pain sensitization in knee-OA subjects with clinical signs of sensitization. However, there is still a paucity of information on the exact exercise mode for greatest beneficial effects in the knee-OA population.

Reduced lower limb muscle strength has repeatedly been suggested as one of the main working mechanisms behind knee-OA symptoms and quadriceps muscle strength is even suggested as a potential mediating factor in future knee joint space narrowing and longitudinal worsening of knee-joint pain. A recent systematic review revealed upper leg muscle strength along with joint proprioception to be two of the most potent mediating factors in symptomatic knee-OA.

In a randomized controlled trial (RCT) design, this study seeks to investigate potential added benefits of supplementing NEMEX and education with focused knee extensor strength training in patients with knee-OA. 90 patients deemed ineligible for knee replacement surgery will be recruited from the ambulatory setting at Naestved Hospital. By random allocation, patients will be recruited to either 12 weeks (twice weekly) of NEMEX and education + focused knee extensor strength training (intervention group) or 12 weeks (twice weekly) of NEMEX and education only (control group).

The main outcome is the change in KOOS-ADL from baseline to 12-week follow-up. Other outcomes include the remaining KOOS subscales, self-reported pain, health status, physical activity and patient satisfaction, knee extensor muscle power and knee extensor maximal contractile strength, pain sensitization, MRI assessed thigh muscle quality and physical function.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic and radiographically confirmed knee-OA who are found not eligible for knee replacement surgery by an orthopaedic surgeon in secondary health care.

Exclusion Criteria:

* Kellgren & Lawrence score of <2 on radiography
* Less than "mild" symptoms (mean score >75 in 0-100 KOOS-ADL)
* Medication: Morphine for pain other than knee-joint pain
* Previous ipsilateral knee arthroplasty
* Rheumatoid arthritis
* Inability to comply with the protocol
* Inadequacy in written and spoken Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Activities of daily living (ADL) | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoints: 6 weeks & 12 months.
  KOOS is a validated and extensively used self-reported outcome measure for people with knee OA. KOOS consists of five subscales, of which the subscale KOOS-ADL will be the primary outcome for this study. KOOS-ADL consists of 17 questions, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). KOOS-ADL has demonstrated a test-retest reliability (ICC) of 0.84-0.94 as well as demonstrating responsiveness to change following physical therapy in knee osteoarthritis.

SECONDARY OUTCOMES:
Muscle power (watt/kg. bodyweight) | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoint: Baseline to 6 weeks.
  Knee extensor muscle power (force times acceleration) will be measured using the Nottingham Power Rig (NPR). The NPR measures the power output in total watt and watt pr. bodyweight in kilograms from a seated push on a flat pedal which is transmitted by a lever and chain to spin a flywheel. The NPR is a safe and reliable method to measure explosive knee extensor muscle power and has been validated as a clinically important measure of muscle function in elderly individuals.
Functional performance (40 m walk & stair-climbs) | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoint: 6 weeks.
  Assessment of functional performance involves time (in seconds) taken to complete a 40 m course at fast walking pace as well as time taken to negotiate 9 steps on a standard step-height stair-way. The tests are part of the recommended functional performance tests in knee osteoarthritis.
Pain medication | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoints: 6 weeks & 12 months.
  Assessment of pain medication intake specific for knee pain. Derived as part of self-reported outcome measure.
KOOS (remaining four subscales) | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoints: 6 weeks & 12 months.
  The four remaining subscales of the validated KOOS questionnaire (see primary outcome for further info on KOOS). The 4 remaining subscales cover: symptoms, pain, sport & recreation and quality of life.
AE (adverse events) & Serious Adverse Events (SAE) | Primary endpoint: From baseline to 12 weeks.. Secondary endpoint: 12 months.
  Continous registration of health issues and injuries. Physiotherapists in charge of the training sessions will monitor potential AE and SAE. Also, during the follow-up visits at week 6 and week 12, the participants will be asked about potential AE's and SAE's using open-probe questions. Finally, the 12 month follow-up will include questions regarding AE's and SAE's during the preceding period from baseline to 12 months.

OTHER OUTCOMES:
Pain sensitization | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoint: 6 weeks.
  Pan sensitization will be assessed through pain pressure cuff algometry (PPCA). The assessment involves placing a pneumatic pressure cuff with automatic inflation around the participant's lower leg. Through four different tests, the participant is asked to rate pain intensity (VAS). The pain scores along with cuff pressure (kPa) is registered. The PPCA is an increasingly used measure of deep-tissue pain sensitization, which allows for multimodal measurements of pain mechanisms in the knee-OA population.
MRI derived muscle quality assessment | Primary endpoint: Change from baseline to 12 weeks.
  In order to assess morphologic changes and changes in muscle quality of the knee extensors, patients will undergo two MRI scans (baseline & follow-up). MRI is considered the gold standard in assessing morphometric muscle changes in humans.
Knee extensor isokinetic dynamometry | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoint: 6 weeks.
  Isokinetic dynamometry will be conducted in order to assess the contractile properties of the knee extensors. The dynamometry assessments will allow for specific strength evaluations and is a validated measure of maximal contractile muscle strength.
Functional performance (chair rise) | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoint: 6 weeks..
  The 30 sec chair-rise (total reps) is part of the recommended functional performance tests in knee OA.
Visual Analog Scale (VAS) | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoint: 6 weeks.
  VAS will be derived for the questions: last 24 hours, last week and after 30 min. of walking.
Widespread Pain Index (WPI) | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoint: 6 weeks & 12 months.
  WPI will be assessed by questions on regional body pain as validated by the American College of Rheumatology.
Numeric Rating Scale (NRS) | Continuous assessments from baseline to 12 weeks.
  NRS will be derived before, during and after each exercise session as well as before and after each testing procedure. The NRS assessments will allow for an evaluation of the effects of exercise and functional activities on self-reported pain ratings.
Physical activity level | Primary endpoint: Change from baseline to 12 weeks. Secondary outcomes: 6 weeks & 12 months.
  Patient reported physical activity levels.
Compliance with exercise | Primary endpoint: 12 weeks..
  The number of exercise sessions that the patient participates in out of the total 24 supervised sessions.
Surgery and other treatments during follow-up | Primary endpoint: 12 weeks. Secondary endpoints: 6 weeks & 12 months.
  Self-reported assessment at baseline, 6 and 12 weeks and at 12 months.
EuroQOL 5 domain | Primary endpoint: Change from baseline to 12 weeks. Secondary endpoints: 6 weeks & 12 months.
  A self-reported outcome measure of health-related quality of life, covering 5 dimensions (movement, personal care, everyday activities, pain/discomfort and anxiety/depression). Is translated and validated for use in a Danish population.
Patient Acceptable Symptom State (PASS) | Primary endpoint: 12 weeks. Secondary endpoint: 6 weeks & 12 months.
  PASS registers how patients perceive their current symptom state. Answered by "yes" or "no" to the question; "When you think of your knee function, will you consider your current condition as satisfying?".
Global Perceived Effect (GPE) | Primary endpoint: 12 weeks. Secondary endpoints: 6 weeks & 12 months.
  GPE registers how patients perceive the effects of the interventions on a 7-point likert scale.
Treatment Failure (TF) | Primary endpoint: 12 weeks. Secondary endpoint: 12 months.
  Only answered by patients answering "no" to PASS. TF registers if the patients perceive the intervention as failed. Answered by "yes" or "no" to the question; "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?".

CONTACTS AND LOCATIONS:
Overall Officials: Pætur M Holm, PT, MSc, Principal Investigator — University of Southern Denmark and Department of Physiotherapy and Occupational Therapy, Naestved-Slagelse-Ringsted Hospitals.; Søren T Skou, PT, PhD, Study Chair — University of Southern Denmark and Naestved-Slagelse-Ringsted Hospitals.; Henrik M Schøder, MD, Study Chair — Naestved Hospital; Mathias Wernbom, PT, PhD, Study Chair — Göteborg University
Locations (1):
- Department of planned Orthopaedic Surgery, Naestved Hospital, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holm PM, Kemnitz J, Bandholm T, Wernbom M, Schroder HM, Skou ST. Muscle Function Tests as Supportive Outcome Measures for Performance-Based and Self-Reported Physical Function in Patients With Knee Osteoarthritis: Exploratory Analysis of Baseline Data From a Randomized Trial. J Strength Cond Res. 2022 Sep 1;36(9):2635-2642. doi: 10.1519/JSC.0000000000003840. Epub 2020 Oct 5. PMID 33021580
- [Derived] Holm PM, Nyberg M, Wernbom M, Schroder HM, Skou ST. Intrarater Reliability and Agreement of Recommended Performance-Based Tests and Common Muscle Function Tests in Knee Osteoarthritis. J Geriatr Phys Ther. 2021 Jul-Sep 01;44(3):144-152. doi: 10.1519/JPT.0000000000000266. PMID 32304510
- [Derived] Holm PM, Schroder HM, Wernbom M, Skou ST. Low-dose strength training in addition to neuromuscular exercise and education in patients with knee osteoarthritis in secondary care - a randomized controlled trial. Osteoarthritis Cartilage. 2020 Jun;28(6):744-754. doi: 10.1016/j.joca.2020.02.839. Epub 2020 Mar 13. PMID 32179197